CLINICAL TRIAL: NCT06798285
Title: Comparision of Retinal Function and Macular Structure After 27G Pars Plana Vitrectomy With Minimal Heads-up Versus Standard Illuminiation in Patients With Idiopthic Epiretinal Membranes
Brief Title: Comparision of Retinal Function and Macular Structure After 27G Pars Plana Vitrectomy With Minimal Illuminiation
Acronym: ERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERM
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria were assigned to groups according to block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (standard): 20 eyes (Active Comparator): Group I (standard): 20 eyes treated using a standard microscope (Hi-R 900, Möller-Wedel Optical GmbH)
  Interventions: Procedure: Pars Plana Vitrectomy Standard
- Group II (3D): 20 eyes (Active Comparator): Group II (3D): 20 eyes treated using the 3D heads-up NGENUITY 3D Visualization System (Alcon Laboratories, Inc.; Fort Worth, TX, USA)
  Interventions: Procedure: Pars Plana Vitrectomy 3D

INTERVENTIONS:
Procedure: Pars Plana Vitrectomy Standard — Group I: PPV with endoillumination set at 3.2 Lm.
  Arms: Group I (standard): 20 eyes
Procedure: Pars Plana Vitrectomy 3D — Group II: PPV with endoillumination set at 0.5 Lm.
  Arms: Group II (3D): 20 eyes

SUMMARY:
Purpose: To analyze the clinical benefits of using the NGENUITY 3D Visualization System in vitreoretinal surgery with low levels of endo-illumination, focusing on functional and structural retinal protection in patients with idiopathic epiretinal membranes (ERM).

Design: Prospective, randomized, comparative study. Methods: Forty pseudophakic patients (29♀, 11♂; age 60-80 years) with ERM underwent 27G pars plana vitrectomy (PPV) and were randomly divided into two groups: Group I (20 eyes, stand-ard microscope [Hi-R 900], endo-illumination 3.2 Lm) and Group II (20 eyes, 3D heads-up NGE-NUITY system, endo-illumination 0.5 Lm). Preoperative and 6-month postoperative evaluations included slit-lamp examination, intraocular pressure (IOP, Pascal tonometer), Distance Best Correct-ed Visual Acuity (DBCVA, logMAR), Central Subfield Thickness (CST), Retinal Nerve Fiber Layer Thickness (RNFL, OCT), Pattern ERG (PERG), multifocal ERG (mfERG), flash ERG (ERG, IS-CEV standards), and retinal sensitivity (HFA macula test). Surgery time, xenon light exposure, ERM/ILM peeling time, fundus autofluorescence (FAF), metamorphopsia incidence, and intra-/postoperative adverse events were analyzed. Results were statistically evaluated (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* DBCVA > 0.1 (Snellen charts)
* Pseudophakia
* ERM without other abnormalities
* Patient's consent to participate in the project with a 6-month follow-up after surgery.

Exclusion Criteria:

* Glaucoma
* AMD
* Systemic diseases known to influence retinal function (e.g., diabetes)
* Psychiatric disorders
* Advanced stages of cardiovascular diseases
* Previous PPV
* High myopia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Bioelectrical Retinal function | 6 months
  The low intensity of endoillumination (0.5 Lm) utilized in PPV with the NGENUITY 3D system may reduce retinal phototoxicity compared to the higher intensity of light (3.2 Lm)

SECONDARY OUTCOMES:
Structural Macula Changes | 6 months
  The low intensity illumination may be a cause of reduced macular structure changes
Changes DBCVA (Distance Best Corrected vision) | 6 months
  The low intensity illumination may be a cause of beter DBCVA after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- II Department of Ophthalmology, Pomeranian Medical University, Szczecin, Zachodnipomorskie, Poland

IPD SHARING:
Plan to Share IPD: No